CLINICAL TRIAL: NCT03578159
Title: Study of Arsha Vidya Chhatralaya Initiative on Health and Functioning of Disadvantaged Tribal Children
Status: Completed | Type: Observational
Sponsor: NMP Medical Research Institute (Other)
Collaborators: Warwick Research Services (Other); Arsha Vidya Tirtha (Other)
Responsible Party: Sponsor
Other Study IDs: NMP/10128
Record Dates: First submitted 2018-06-24; First posted 2018-07-06 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-06

CONDITIONS: Physical Disorder; Mental Health Wellness; Social Function Disorder, Childhood or Adolescent; Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Arsha Vidya Chhatralaya: Chhatralaya is residential setting for children 8 to 16 years old. It provides residence,food and education opportunities along with regular practice of Yoga, Spiritual sessions and vedic practices to learn and follow.
  Interventions: Other: Chhatralaya

INTERVENTIONS:
Other: Chhatralaya — Chhatralaya, home for children provide living resources along with spiritual practices.

SUMMARY:
India's poor tribal communities have far worse health and social indicators than the general population. Most tribal people live in remote forested or desert areas where illiteracy, trying physical environments, malnutrition, inadequate access to potable water, and lack of personal hygiene and sanitation make them more vulnerable to disease.The aim of Chhatralaya initiatives taken by Arsha Vidya, Jaipur was to address the exclusion of the socially and economically disadvantaged children of the tribes and to provide a fair opportunity to all.

ELIGIBILITY:
Inclusion Criteria:

* Children selected from Udaipur tribal areas as lacking parental care and basic services;
* Children living in Udaipur tribal areas;
* Children from 8 years to 16 years of age

Exclusion Criteria:

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children selected from Udaipur tribal areas, Rajasthan, India
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-06-08 (Actual)

PRIMARY OUTCOMES:
Physical health and wellbeing | Change from baseline to one year
  Measured by MacArthur Health and Behavior Questionnaire
Mental Health and wellbeing | Change from baseline to one year
  Measured by MacArthur Health and Behavior Questionnaire
Social functioning | Change from baseline to one year
  Measured by MacArthur Health and Behavior Questionnaire
Academic functioning | Change from baseline to one year
  Measured by MacArthur Health and Behavior Questionnaire

SECONDARY OUTCOMES:
Weight | Change from baseline to one year
  child's weight was measured by using a calibrated electronic weighing scale
Prevalence of acute child malnutrition | Change from baseline to one year
  To calculate WHZ scores the 2006 WHO growth reference was used

CONTACTS AND LOCATIONS:
Overall Officials: Brahmaparananda Saraswati, Study Chair — Arsha Vidya Tirtha; Neha Sharma, PhD, Study Director — Warwick Research Servives, UK; Puneet Sharma, Principal Investigator — NMP Medical Research Institute
Locations (1):
- Arsha Vidya Chhatralaya,, Jaipur, Rajasthan, India

IPD SHARING:
Plan to Share IPD: Undecided